CLINICAL TRIAL: NCT01135433
Title: A Phase 3 Study to Assess the Efficacy and Safety of ASP1941 in Combination With Metformin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Alone
Brief Title: A Study to Assess the Efficacy and Safety of ASP1941 in Combination With Metformin in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-0106
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus; Metformin; ASP1941
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP group (Experimental): ASP1941 and metformin
  Interventions: Drug: ipragliflozin; Drug: metformin
- Placebo group (Placebo Comparator): placebo and metformin
  Interventions: Drug: Placebo; Drug: metformin

INTERVENTIONS:
Drug: ipragliflozin — oral
  Other Names: ASP1941
  Arms: ASP group
Drug: Placebo — oral
  Arms: Placebo group
Drug: metformin — oral
  Other Names: Metgluco; Melbin; Glycoran

SUMMARY:
This study is to evaluate the efficacy and safety after concomitant administration of ASP1941 and metformin in patients with diabetes mellitus.

DETAILED DESCRIPTION:
This study is to evaluate the efficacy (HbA1c change from baseline) and safety of ASP1941 in combination with metformin in subjects with type 2 diabetes mellitus (T2DM) who have inadequate glycemic control with metformin alone. The effects of ASP1941 are compared with those of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients receiving with metformin mono-therapy for at least 6 weeks
* HbA1c value between 7.0 and 9.5%
* Body Mass Index (BMI) 20.0 - 45.0 kg/m2

Exclusion Criteria:

* Type 1 diabetes mellitus patients
* Serum creatinine > upper limit of normal
* Estimated GFR < 60ml/min/1.73m2
* Proteinuria (albumin/creatinine ratio > 300mg/g)
* Dysuria and/or urinary tract infection, genital infection
* Significant renal, hepatic or cardiovascular diseases
* Severe gastrointestinal diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-05-15 (Actual); Primary Completion 2011-11-28 (Actual); Study Completion 2011-11-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline and for 24 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose | Baseline and for 24 weeks
Change from baseline in fasting serum insulin | Baseline and for 24 weeks
Safety as reflected by adverse events, routine safety laboratories, vital signs, physical examinations and 12-lead electrocardiograms (ECGs) | for 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=100